CLINICAL TRIAL: NCT01151137
Title: A Randomized, Double Blind, Placebo Controlled, Parallel Group Trial for Assessing the Clinical Benefit of Dronedarone 400mg BID on Top of Standard Therapy in Patients With Permanent Atrial Fibrillation and Additional Risk Factors
Brief Title: Permanent Atrial fibriLLAtion Outcome Study Using Dronedarone on Top of Standard Therapy
Acronym: PALLAS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped because of safety concerns
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EFC11405; 2010-019791-73 (EudraCT Number); U1111-1116-5566 (Other: UTN)
Record Dates: First submitted 2010-06-22; First posted 2010-06-25 (Estimated); Results first posted 2012-10-26 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dronedarone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Dronedarone (Experimental): Dronedarone 400 mg twice a day until the CSED
  Interventions: Drug: Dronedarone
- placebo (Placebo Comparator): Placebo (for Dronedarone) twice a day until the CSED
  Interventions: Drug: Placebo (for Dronedarone)

INTERVENTIONS:
Drug: Dronedarone — Film-coated tablet
  Oral administration under fed conditions (during breakfast and dinner)
  Other Names: MULTAQ; SR33589
  Arms: Dronedarone
Drug: Placebo (for Dronedarone) — film-coated tablet strictly identical in appearance
  Oral administration under fed conditions (during breakfast and dinner)
  Arms: placebo

SUMMARY:
Primary Objective:

* Demonstrate the efficacy of Dronedarone in preventing major cardiovascular events (stroke, systemic arterial embolism, myocardial infarction or cardiovascular death) or unplanned cardiovascular hospitalization or death from any cause in patients with permanent Atrial Fibrillation [AF] and additional risk factors

Secondary Objective:

* Demonstrate the efficacy of Dronedarone in preventing cardiovascular death

This was an event-driven study where a common study end date [CSED] was to be determined by Steering Committee based on the number of events (stroke, systemic arterial embolism, myocardial infarction or cardiovascular death).

DETAILED DESCRIPTION:
The study period per participant was variable depending on the enrollment in the study.

A final follow-up visit had to occur within 1 month after the CSED.

ELIGIBILITY:
Inclusion criteria:

* Permanent AF defined by the presence of all of the following criteria:

  * Availability of one 12-lead ECG not more than 14 days prior to randomization showing that the patient is in AF or atrial flutter;
  * Availability of documentation (including either rhythm strips or medical report of the rhythm) showing that the patient was in AF or atrial flutter at least 6 months prior to randomization;
  * No evidence of sinus rhythm in the period between these two documentations of AF;
  * Decision of the patient and physician to allow AF to continue without further efforts to restore sinus rhythm.
* At least one of the following risk criteria:

  * Coronary artery disease;
  * Prior stroke or Transient Ischemic Attack [TIA];
  * Symptomatic heart failure;
  * Left ventricular ejection fraction [LVEF] less or equal to 0.40;
  * Peripheral arterial occlusive disease;
  * Aged 75 years or older with both hypertension and diabetes mellitus.

Exclusion criteria:

* Paroxysmal AF;
* Persistent AF without a decision to allow AF to continue without further efforts to restore sinus rhythm;
* Heart failure of New-York Heart Association [NYHA] class IV or recent unstable NYHA class III.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 3236 (Actual)
Dates: Start 2010-07; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (37):
- Sanofi-Aventis Administrative Office, Bridgewater, New Jersey, United States
- Sanofi-Aventis Administrative Office, Buenos Aires, Argentina
- Sanofi-Aventis Administrative Office, Macquarie Park, Australia
- Sanofi-Aventis Administrative Office, Vienna, Austria
- Sanofi-Aventis Administrative Office, Diegem, Belgium
- Sanofi-Aventis Administrative Office, São Paulo, Brazil
- Sanofi-Aventis Administrative Office, Sofia, Bulgaria
- Sanofi-Aventis Administrative Office, Laval, Canada
- Sanofi-Aventis Administrative Office, Providencia Santiago, Chile
- Sanofi-Aventis Administrative Office, Prague, Czechia
- Sanofi-Aventis Administrative Office, Hørsholm, Denmark
- Sanofi-Aventis Administrative Office, Helsinki, Finland
- Sanofi-Aventis Administrative Office, Paris, France
- Sanofi-Aventis Administrative Office, Frankfurt, Germany
- Sanofi-Aventis Administrative Office, Kallithea, Greece
- Sanofi-Aventis Administrative Office, Hong Kong, Hong Kong
- Sanofi-Aventis Administrative Office, Budapest, Hungary
- Sanofi-Aventis Administrative Office, Netanya, Israel
- Sanofi-Aventis Administrative Office, Milan, Italy
- Sanofi-Aventis Administrative Office, Kuala Lumpur, Malaysia
- Sanofi-Aventis Administrative Office, Col. Coyoacan, Mexico
- Sanofi-Aventis Administrative Office, Gouda, Netherlands
- Sanofi-Aventis Administrative Office, Auckland, New Zealand
- Sanofi-Aventis Administrative Office, Lysaker, Norway
- Sanofi-Aventis Administrative Office, Warsaw, Poland
- Sanofi-Aventis Administrative Office, Bucharest, Romania
- Sanofi-Aventis Administrative Office, Moscow, Russia
- Sanofi-Aventis Administrative Office, Singapore, Singapore
- Sanofi-Aventis Administrative Office, Bratislava, Slovakia
- Sanofi-Aventis Administrative Office, Gauteng, South Africa
- Sanofi-Aventis Administrative Office, Seoul, South Korea
- Sanofi-Aventis Administrative Office, Barcelona, Spain
- Sanofi-Aventis Administrative Office, Bromma, Sweden
- Sanofi-Aventis Administrative Office, Geneva, Switzerland
- Sanofi-Aventis Administrative Office, Taipei, Taiwan
- Sanofi-Aventis Administrative Office, Kiev, Ukraine
- Sanofi-Aventis Administrative Office, Guildford Surrey, United Kingdom

REFERENCES:
- [Result] Connolly SJ, Camm AJ, Halperin JL, Joyner C, Alings M, Amerena J, Atar D, Avezum A, Blomstrom P, Borggrefe M, Budaj A, Chen SA, Ching CK, Commerford P, Dans A, Davy JM, Delacretaz E, Di Pasquale G, Diaz R, Dorian P, Flaker G, Golitsyn S, Gonzalez-Hermosillo A, Granger CB, Heidbuchel H, Kautzner J, Kim JS, Lanas F, Lewis BS, Merino JL, Morillo C, Murin J, Narasimhan C, Paolasso E, Parkhomenko A, Peters NS, Sim KH, Stiles MK, Tanomsup S, Toivonen L, Tomcsanyi J, Torp-Pedersen C, Tse HF, Vardas P, Vinereanu D, Xavier D, Zhu J, Zhu JR, Baret-Cormel L, Weinling E, Staiger C, Yusuf S, Chrolavicius S, Afzal R, Hohnloser SH; PALLAS Investigators. Dronedarone in high-risk permanent atrial fibrillation. N Engl J Med. 2011 Dec 15;365(24):2268-76. doi: 10.1056/NEJMoa1109867. Epub 2011 Nov 14. PMID 22082198
- [Derived] Hohnloser SH, Halperin JL, Camm AJ, Gao P, Radzik D, Connolly SJ; PALLAS investigators. Interaction between digoxin and dronedarone in the PALLAS trial. Circ Arrhythm Electrophysiol. 2014 Dec;7(6):1019-25. doi: 10.1161/CIRCEP.114.002046. Epub 2014 Nov 6. PMID 25378467

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment initiated in July 2010 was discontinued on July 6, 2011 upon recommendations of the Data Monitoring Committee due to an increased number of observed cardiovascular events in the Dronedarone group. The common study end date [CSED] was defined as July 15, 2011.
  At that time 494 sites in 37 countries had enrolled at least one patient.
Pre-assignment Details: Assignment to groups was done centrally using an Interactive Voice Response System [IVRS] or an Interactive Web Response System [IWRS] in a 1:1 ratio.
  A total of 3236 participants were randomized at 489 sites (instead of 10800 as initially planned). The median duration of their participation in the study was 3.5 months.
Groups:
- Placebo: Placebo twice daily until the CSED (median treatment duration of 87.5 days)
- Dronedarone: Dronedarone 400 mg twice daily until the CSED (median treatment duration of 74 days)
Period: Overall Study
Arm/Group | Placebo | Dronedarone
Started | 1617 | 1619
Treated | 1610 (One participant randomized to the placebo group received Dronedarone for 7 days by mistake) | 1613
Discontinued Treatment | 171 | 342
Completed | 1601 | 1591
Not Completed | 16 | 28
Not completed — Death | 15 | 27
Not completed — Lost to Follow-up | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Dronedarone | Total
Number analyzed (Participants) | 1617 | 1619 | 3236
Age Continuous [Mean (Standard Deviation); unit: years] | 75.0 (5.9) | 75.0 (5.9) | 75.0 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 577 | 568 | 1145
  Male | 1040 | 1051 | 2091
Region of Enrollment [Number; unit: participants] — Regions were defined as follows:
  * North America: Canada, United States
  * South America: Argentina, Brazil, Chile, Mexico
  * Western Europe: Austria, Belgium, Denmark, Finland, France, Germany, Greece, Italy, Netherlands, Norway, Spain, Sweden, Switzerland, United Kingdom
  * Eastern Europe: Bulgaria, Czech Republic, Hungary, Poland, Romania, Russian Federation, Slovakia, Ukraine Asia: Hong Kong, Republic of Korea, Malaysia, Singapore, Taiwan Rest of the World: Australia, Israel, New zealand, South Africa
  participants
    North America | 281 | 266 | 547
    South America | 227 | 236 | 463
    Western Europe | 459 | 475 | 934
    Eastern Europe | 495 | 488 | 983
    Asia | 53 | 47 | 100
    Rest of the word | 102 | 107 | 209
Permanent atrial fibrillation [AF] history [Number; unit: participants]
  6 months to 2 years | 490 | 498 | 988
  > 2 years | 1124 | 1119 | 2243
  Unknown | 3 | 2 | 5
CHADS2 Score [Number; unit: participants] — CHADS2 is a risk-prediction score ranging from 0 to 6 used estimate Stroke Risk in Atrial Fibrillation patients.
  CHADS2 score is obtained by adding together the points that correspond to the conditions that are present:
  * C: Congestive Heart Failure history: 1 point
  * H: Hypertension history: 1 point
  * A: Age ≥75 years: 1 point
  * D: Diabetes Mellitus history: 1 point
  * S: Stroke symptoms previously or Transient Ischemic Attack [TIA]: 2 points
  participants
    < 2 | 172 | 191 | 363
    ≥ 2 | 1444 | 1427 | 2871
    Unavailable | 1 | 1 | 2
New York Heart Association [NYHA] class [Number; unit: participants] — NYHA classification is a functional classification that places the patient in one of 4 categories, based on how much he/she is limited during physical activity:
  * Class I: no limitation of activities; the patient suffers no symptoms from ordinary activities.
  * Class II: slight, mild limitation of activity; the patient is comfortable with rest or with mild exertion.
  * Class III: marked limitation of activity; the patient is comfortable only at rest.
  * Class IV: complete rest, confined to bed or chair; any physical activity brings on discomfort and symptoms occur at rest.
  participants
    No congestive heart failure [CHF] | 535 | 512 | 1047
    NYHA Class I | 209 | 234 | 443
    NYHA Class II | 749 | 732 | 1481
    NYHA Class III | 124 | 141 | 265

OUTCOME MEASURES:

1. Primary Outcome: Overview of the Two Co-primary Outcomes
Description: First co-primary outcome was defined as the first event among stroke, systemic arterial embolism, Myocardial Infarctions [MI], or cardiovascular death.
  Second co-primary outcome was defined as the first event among unscheduled cardiovascular hospitalization or death from any cause.
  Both co-primary outcomes were determined based on the central review and adjudication by a blinded Adjudication Committee of all reported deaths (from any cause), MI, systemic arterial embolisms, strokes, Transient Ischemic Attacks [TIA], Heart Failure hospitalization and unplanned hospitalisations for cardiovascular cause.
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population: All randomized participants considered in the treatment group to which they were randomized regardless of the treatment they actually received
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
participants
  First co-primary endpoint | 19 | 43
  Second co-primary endpoint | 67 | 127

2. Primary Outcome: Time to First Co-primary Outcome (Cumulative Incidence Function)
Description: Time to first co-primary outcome was defined as the time from randomization to the first event among stroke, systemic arterial embolism, MI or cardiovascular death.
  Cumulative incidence function in each treatment group was calculated using non-parametric Kaplan-Meier estimate.
  95% confidence interval was computed at each time-point using Greenwood's variance estimation.
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population as previously defined
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
proportion of participants
  Cumulative incidence at 14 days | 0.002 [0.000 to 0.004] | 0.009 [0.005 to 0.014]
  Cumulative incidence at 30 days | 0.003 [0.000 to 0.006] | 0.013 [0.008 to 0.019]
  Cumulative incidence at 90 days | 0.007 [0.003 to 0.012] | 0.021 [0.014 to 0.029]
  Cumulative incidence at 180 days | 0.013 [0.006 to 0.021] | 0.042 [0.028 to 0.056]
  Cumulative incidence at 270 days | 0.038 [0.012 to 0.064] | 0.045 [0.030 to 0.061]
  Cumulative incidence at 360 days | 0.038 [0.012 to 0.064] | 0.045 [0.030 to 0.061]
Statistical Analysis 1: Comparison: Placebo vs Dronedarone; As a consequence of the early termination of the study, the analysis was performed for information only without any adjustment; Test type: Superiority or Other; p = 0.0019, Log Rank — A priori threshold for statistical significance: 0.05; 2-sided Log-rank's asymptotic test; Hazard Ratio (HR) = 2.294, 95% CI 2-sided [1.337 to 3.936] — Hazard ratio (HR) of Dronedarone versus placebo for stroke, systemic arterial embolism, myocardial infarction or cardiovascular death HR and confidence interval were estimated using Cox regression model with treatment group as the only factor

3. Primary Outcome: Time to Second Co-primary Outcome (Cumulative Incidence Function)
Description: Time to second co-primary outcome was defined as the time from randomization to the first event among unscheduled cardiovascular hospitalization or death from any cause.
  Cumulative incidence function in each treatment group was calculated using non-parametric Kaplan-Meier estimate.
  95% confidence interval was computed at each time-point using Greenwood's variance estimation.
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population as previously defined
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
proportion of participants
  Cumulative incidence at 14 days | 0.005 [0.002 to 0.008] | 0.020 [0.013 to 0.027]
  Cumulative incidence at 30 days | 0.014 [0.008 to 0.020] | 0.034 [0.025 to 0.043]
  Cumulative incidence at 90 days | 0.033 [0.023 to 0.042] | 0.069 [0.055 to 0.083]
  Cumulative incidence at 180 days | 0.059 [0.043 to 0.075] | 0.110 [0.089 to 0.130]
  Cumulative incidence at 270 days | 0.099 [0.062 to 0.137] | 0.137 [0.107 to 0.167]
  Cumulative incidence at 360 days | 0.099 [0.062 to 0.137] | 0.137 [0.107 to 0.167]
Statistical Analysis 1: Comparison: Placebo vs Dronedarone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Log Rank — A priori threshold for statistical significance: 0.05; 2-sided Log-rank's asymptotic test; Hazard Ratio (HR) = 1.947, 95% CI 2-sided [1.448 to 2.617] — Hazard ratio (HR) of Dronedarone versus placebo for unscheduled cardiovascular hospitalization or death from any cause HR and confidence interval were estimated using Cox regression model with treatment group as the only factor

4. Secondary Outcome: Deaths
Description: Deaths were classified according to the primary cause of death.
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population as previously defined
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
participants
  Any death | 13 | 25
  - Cardiovascular death | 10 | 21
  --- Cardiac arrhythmic death | 4 | 13

5. Secondary Outcome: Time to Cardiovascular Death (Cumulative Incidence Function)
Description: Time to cardiovascular death was defined as the time from randomization to the death.
  Cumulative incidence function in each treatment group was calculated using non-parametric Kaplan-Meier estimate.
  95% confidence interval was computed at each time-point using Greenwood's variance estimation.
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population as previously defined
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
proportion of participants
  Cumulative incidence at 14 days | 0.001 [0.000 to 0.003] | 0.003 [0.000 to 0.006]
  Cumulative incidence at 30 days | 0.003 [0.000 to 0.006] | 0.005 [0.002 to 0.009]
  Cumulative incidence at 90 days | 0.004 [0.001 to 0.007] | 0.008 [0.003 to 0.012]
  Cumulative incidence at 180 days | 0.004 [0.001 to 0.007] | 0.022 [0.012 to 0.033]
  Cumulative incidence at 270 days | 0.027 [0.001 to 0.052] | 0.026 [0.013 to 0.038]
  Cumulative incidence at 360 days | 0.027 [0.001 to 0.052] | 0.026 [0.013 to 0.038]
Statistical Analysis 1: Comparison: Placebo vs Dronedarone; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0460, Log Rank — A priori threshold for statistical significance: 0.05; 2-sided Log-rank's asymptotic test; Hazard Ratio (HR) = 2.115, 95% CI 2-sided [0.996 to 4.490] — Hazard ratio (HR) of Dronedarone versus placebo for cardiovascular death HR and confidence interval were estimated using Cox regression model with treatment group as the only factor

6. Other Pre Specified Outcome: Overview of Cardiovascular Events
Time Frame: From randomization up to the CSED which occurred at study termination (maximum follow-up of 1 year)
Population: Intent-to-treat population as previously defined
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1617 | 1619
participants
  MI or unstable angina pectoris | 8 | 15
  - MI | 2 | 3
  Stroke | 10 | 23
  - Ischemic stroke | 9 | 18
  Systemic arterial embolism | 0 | 1
  Episode of heart failure | 55 | 115
  - Hospitalization due to heart failure | 24 | 43
  Unplanned hospitalization for cardiovascular cause | 59 | 113

7. Other Pre Specified Outcome: Overview of Adverse Events [AE]
Description: AE are any unfavorable and unintended sign, symptom, syndrome, or illness observed by the investigator or reported by the participant during the study.
Time Frame: from first study drug intake up to 10 days after the last study drug intake
Population: Safety population: all randomized and treated participants. Participants were considered according to the treatment actually received. Consequently the participant randomized to the placebo group who received Dronedarone was included in the Dronedarone group.
Measure: Number; unit: participants
Arm/Group | Placebo | Dronedarone
Number analyzed (Participants) | 1609 | 1614
participants
  Any AE | 600 | 797
  - Any serious AE | 77 | 113
  - Any AE leading to death | 0 | 4
  - Any AE leading to treatment discontinuation | 80 | 212
  - Any AE leading to hospitalization | 71 | 95

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected regardless of seriousness or relationship to the drug, spanning from signature of the Informed Consent Form up to the last visit.
Description: The analysis included all randomized participants who received at least one dose of study drug and all AE that developed or worsened from randomization up to 10 days after last study drug intake.
  Participants were considered according to the treatment actually received regardless the amount of treatment administered.
Arm/Group | Placebo | Dronedarone
Serious Adverse Events (participants affected / at risk) | 77/1609 | 113/1614
Other Adverse Events (participants affected / at risk) | 38/1609 | 100/1614
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1609) | Dronedarone (N=1614)
Bronchitis (Infections and infestations) | 1 | 2
Urinary tract infection (Infections and infestations) | 2 | 2
Pneumonia (Infections and infestations) | 9 | 10
Gastroenteritis (Infections and infestations) | 0 | 3
Cellulitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 2 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1
Escherichia sepsis (Infections and infestations) | 0 | 1
Lobar pneumonia (Infections and infestations) | 1 | 1
Otitis media chronic (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 1
Arthritis bacterial (Infections and infestations) | 0 | 1
Intervertebral discitis (Infections and infestations) | 0 | 1
Clostridial infection (Infections and infestations) | 0 | 1
Fungal peritonitis (Infections and infestations) | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 2 | 0
Gangrene (Infections and infestations) | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0
Prostate cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Myeloproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 0
Gout (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 2 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0
Electrolyte depletion (Metabolism and nutrition disorders) | 0 | 1
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Diabetic foot (Metabolism and nutrition disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 0 | 1
Delirium (Psychiatric disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 2 | 1
Presyncope (Nervous system disorders) | 0 | 2
Diabetic neuropathy (Nervous system disorders) | 0 | 1
Encephalitis (Nervous system disorders) | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Optic ischaemic neuropathy (Eye disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Hypovolaemic shock (Vascular disorders) | 0 | 1
Orthostatic hypotension (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Idiopathic pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Colitis (Gastrointestinal disorders) | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0
Subileus (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Ileitis (Gastrointestinal disorders) | 0 | 1
Inguinal hernia (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Abdominal wall haematoma (Gastrointestinal disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 2
Cholelithiasis (Hepatobiliary disorders) | 2 | 2
Acute hepatic failure (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 1
Hepatic congestion (Hepatobiliary disorders) | 0 | 1
Hepatitis (Hepatobiliary disorders) | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer haemorrhage (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 2 | 3
Renal failure acute (Renal and urinary disorders) | 1 | 8
Haematuria (Renal and urinary disorders) | 1 | 2
Renal failure chronic (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 1
Acquired hydrocele (Reproductive system and breast disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 1 | 0
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0
Oedema peripheral (General disorders) | 1 | 0
Chest pain (General disorders) | 0 | 2
Non-cardiac chest pain (General disorders) | 1 | 1
Generalised oedema (General disorders) | 1 | 0
Blood creatinine increased (Investigations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Hepatic enzyme increased (Investigations) | 1 | 5
Fall (Injury, poisoning and procedural complications) | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Multiple fractures (Injury, poisoning and procedural complications) | 0 | 1
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 | 1
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Eventration procedure (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=1609) | Dronedarone (N=1614)
Diarrhoea (Gastrointestinal disorders) | 38 | 100

LIMITATIONS AND CAVEATS:
Given that the study was prematurely discontinued after 3236 patients were randomized (30% of the initial planned number), p-values were provided for information without any adjustment for multiplicity.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months after trial completion, the investigator can present or publish trial results. A copy is submitted to the sponsor for review and comment at least 30 days in advance of any presentation or submission for publication.

The sponsor can require to delay the communication for a period not exceeding 90 days to allow for filing a patent application or such other measures as sponsor deems appropriate to establish and preserve its proprietary rights.